CLINICAL TRIAL: NCT00557414
Title: Serial Changes of sTREM-1 Levels in Patients With Acute Respiratory Distress Syndrome
Brief Title: Serial Changes of Soluble Triggering Receptor Expressed on Myeloid Cells-1 (sTREM-1) Levels in Patients With Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chao-Chi Ho, National Taiwan University Hospital
Other Study IDs: 200709060R
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Last update posted 2008-05-13 (Estimated); Status verified 2008-05

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: acute respiratory distress syndrome; soluble triggering receptor expressed on myeloid cells-1; prognosis
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine the impact of the serum soluble triggering receptor expressed on myeloid cells-1 (sTREM-1) on etiology and prognosis of acute respiratory distress syndrome (ARDS)

DETAILED DESCRIPTION:
The triggering receptor expressed on myeloid cells-1 (TREM-1), a member of the immunoglobulin superfamily, is upregulated on phagocytic cells in the presence of bacteria or fungi infection and weakly expressed in samples from patients with noninfectious inflammatory disorders. In addition, TREM-1 is shed from the membrane of activated phagocytes and can be found in a soluble form (sTREM-1) in body fluids. The level and serial change of a serum sTREM-1 from cirtical ill patients has been shown to be a good diagnostic and prognostic indicator of ventilation associated pneumonia (VAP) and severe sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill clinical diagnosis of ARDS
* Require mechanical ventilation support

Exclusion Criteria:

* Pregnant
* Immunocompromised

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted into ICU of a medical center in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2007-10; Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
all cause mortality | 28 days
Septic or non-septic etiology | At enrollment

SECONDARY OUTCOMES:
CRP, lactate, WBC count, APACHE II score, LIS, SOFA score | At enrollment
IL-1 beta, IL-8, TNF-alpha | serial follow up at Day 1, 3, 5, 7, 14

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Chi Ho, Principal Investigator — Department of Internal Medicine and Emergency Medicine, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan